CLINICAL TRIAL: NCT07071519
Title: A Phase 3, Multi-Center Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Risankizumab With Open-Label Induction, Randomized Double-Blind Maintenance, and Open-Label Long-Term Extension Periods in Pediatric Subjects (2 to < 18 Years of Age) With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Learn More About How Risankizumab Works in Young Participants With Ulcerative Colitis
Acronym: MIGHTY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: M19-751
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
Keywords: risankizumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- PK Cohort 1: SS1 (Experimental): Cohort 1 will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All participants who complete SS1 are eligible to enter SS2
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS2 Dose A (Experimental): Cohort 1 will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long term extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS2 Dose B (Experimental): Cohort 1 will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long term extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS3 Dose A (Experimental): Cohort 1 will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS3 Dose B (Experimental): Cohort 1 will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS1 (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All subjects who complete SS1 are eligible to enter SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS2 Dose A (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long-term extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS2 Dose B (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long-term extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS3 Dose A (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS3 Dose B (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS1 (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All participants who complete SS1 are eligible to enter SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS2 Dose A (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long term extension SS3.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS2 Dose B (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long term extension SS3.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS3 Dose A (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS3 Dose B (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab intravenous (IV) infusion
  Other Names: ABBV-066
  Arms: Expansion Cohort 3: SS1; PK Cohort 1: SS1; PK Cohort 2: SS1
Drug: Risankizumab — Risankizumab subcutaneous (SC) injection
  Other Names: ABBV-066
  Arms: Expansion Cohort 3: SS2 Dose A; Expansion Cohort 3: SS2 Dose B; Expansion Cohort 3: SS3 Dose A; Expansion Cohort 3: SS3 Dose B; PK Cohort 1: SS2 Dose A; PK Cohort 1: SS2 Dose B; PK Cohort 1: SS3 Dose A; PK Cohort 1: SS3 Dose B; PK Cohort 2: SS2 Dose A; PK Cohort 2: SS2 Dose B; PK Cohort 2: SS3 Dose A; PK Cohort 2: SS3 Dose B

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). This study will assess how Risankizumab moves through the body as well as how safe and effective it is in treating pediatric participants with moderate to severely active UC. Adverse events and change in disease activity will be assessed.

Risankizumab is an approved medication for moderate to severe UC in multiple countries and is being developed for the treatment of UC in pediatrics. This study is comprised of 3 cohorts that may participate in 3 substudies (SS). Cohort 1 will enroll participants with ages from 6 to less than 18 years. Cohort 2 will enroll participants with ages from 2 to less than 6 years. Cohort 3 will enroll participants with ages from 2 to less than 18 years. SS1 is an open-label induction period where participants will receive a weight-based induction regimen of risankizumab. SS2 is a double-blind maintenance period where participants will be randomized to receive 1 of 2 doses of weight-based maintenance regimen of risankizumab. SS3 is an open-label extension period where participants will receive risankizumab based off of their response in SS2. Around 120 pediatric participants with UC will be enrolled at around 80 sites worldwide.

Participants in SS1 will receive risankizumab intravenously during the 12-week induction period. Participants in SS2 will receive risankizumab subcutaneously during the 52-week randomized maintenance period. Participants in SS3 will receive risankizumab subcutaneously during the 208-week open label period. Participants will be followed-up for approximately 140 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis (UC) with an modified Mayo Score (mMS) of 5 to 9 points and endoscopic subscore of 2 to 3 (confirmed by central reader).
* Demonstrated intolerance or inadequate response (IR) to one or more of the following categories of drugs:

aminosalicylates (except in countries where failure of this drug class is not sufficient for eligibility), oral locally acting corticosteroids, systemic steroids (prednisone or equivalent), immunomodulators (IMMs), and/or biologic therapies, as outlined in the protocol.

- Subjects must have a documented history of UC for at least 3 months prior to Baseline, confirmed by colonoscopy during the screening period, with exclusion of current infection, colonic dysplasia and/or malignancy. Documentation of pathology results consistent with the diagnosis of UC must be available.

Exclusion Criteria:

* Participants who have had a major surgery performed within 12 weeks prior to Baseline or planned during the conduct of the study (e.g., inguinal hernia repair, cholecystectomy, intestinal resection).
* Participants who have concurrent clinically significant medical conditions other than the indication being studied or any other reason that the investigator determines would interfere with the subject's participation in this study, would make the subject an unsuitable candidate to receive study treatment, or would put the subject at risk by participating in the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2034-07 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
PK Lead-In Cohort 1: Maximum Observed Serum Concentration (Cmax) | At Week 64
  Maximum observed plasma concentration (Cmax)
PK Lead-In Cohort 2: Maximum Observed Serum Concentration (Cmax) | At Week 64
  Maximum observed plasma concentration (Cmax)
PK Lead-In Cohort 1: Time to Maximum Serum Concentration (Tmax) | At Week 64
  Time to maximum plasma concentration (Tmax)
PK Lead-In Cohort 2: Time to Maximum Serum Concentration (Tmax) | At Week 64
  Time to maximum plasma concentration (Tmax)
PK Lead-In Cohort 1: Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) | At Week 64
  Area under the serum concentration-time curve over the dosing interval (AUCtau)
PK Lead-In Cohort 2: Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) | At Week 64
  Area under the serum concentration-time curve over the dosing interval (AUCtau)
Expansion Cohort 3: Achievement of Clinical Remission per Modified Mayo Score (mMS) Among Week 12 Clinical Responders per mMS | At Week 64
  Clinical remission on the mMS is defined as defined as Stool Frequency Subscore (SFS) ≤ 1 and not greater than Baseline, Rectal Bleeding Subscore (RBS) = 0, and Mayo Endoscopic Subscore (MES) ≤ 1
Number of Participants With Adverse Events | Up to 292 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related

SECONDARY OUTCOMES:
PK Lead-In Cohort 1: Achievement of clinical remission per mMS among Week 12 responders per mMS | At Week 64
  Clinical remission on the mMS is defined as defined as Stool Frequency Subscore (SFS) ≤ 1 and not greater than Baseline, Rectal Bleeding Subscore (RBS) = 0, and Mayo Endoscopic Subscore (MES) ≤ 1
PK Lead-In Cohort 2: Achievement of clinical remission per mMS among Week 12 responders per mMS | At Week 64
  Clinical remission on the mMS is defined as defined as Stool Frequency Subscore (SFS) ≤ 1 and not greater than Baseline, Rectal Bleeding Subscore (RBS) = 0, and Mayo Endoscopic Subscore (MES) ≤ 1
PK Lead-In Cohort 1: Achievement of clinical remission per mMS | At Week 12
  Clinical remission on the mMS is defined as Stool Frequency Subscore (SFS) ≤ 1 and not greater than Baseline, Rectal Bleeding Subscore (RBS) = 0, and Mayo Endoscopic Subscore (MES) ≤ 1
PK Lead-In Cohort 2: Achievement of clinical remission per mMS | At Week 12
  Clinical remission on the mMS is defined as Stool Frequency Subscore (SFS) ≤ 1 and not greater than Baseline, Rectal Bleeding Subscore (RBS) = 0, and Mayo Endoscopic Subscore (MES) ≤ 1
PK Lead-In Cohort 1: Achievement of clinical response per mMS | At Week 12
  Clinical response per mMS is defined as decrease in mMS by ≥ 2 points and ≥ 30% from Baseline with a decrease in Rectal Bleeding Subscore (RBS) of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 2: Achievement of clinical response per mMS | At Week 12
  Clinical response per mMS is defined as decrease in mMS by ≥ 2 points and ≥ 30% from Baseline with a decrease in Rectal Bleeding Subscore (RBS) of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 1: Achievement of endoscopic improvement | At Week 12
  Endoscopic improvement defined as MES ≤ 1
PK Lead-In Cohort 2: Achievement of endoscopic improvement | At Week 12
  Endoscopic improvement defined as MES ≤ 1
PK Lead-In Cohort 1: Symptomatic response per partial mMS | At Week 12
  Symptomatic response per partial mMS is defined as decrease in partial mMS by ≥ 1 points and ≥ 30% from Baseline with decrease in RBS of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 2: Symptomatic response per partial mMS | At Week 12
  Symptomatic response per partial mMS is defined as decrease in partial mMS by ≥ 1 points and ≥ 30% from Baseline with decrease in RBS of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 1: Achievement of clinical response per mMS among Week 12 responders per mMS | At Week 64
  Clinical response per mMS is defined as decrease in mMS by ≥ 2 points and ≥ 30% from Baseline with a decrease in Rectal Bleeding Subscore (RBS) of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 2: Achievement of clinical response per mMS among Week 12 responders per mMS | At Week 64
  Clinical response per mMS is defined as decrease in mMS by ≥ 2 points and ≥ 30% from Baseline with a decrease in Rectal Bleeding Subscore (RBS) of ≥ 1 or an absolute RBS of 0 or 1.
PK Lead-In Cohort 1: Achievement of endoscopic improvement among Week 12 responders per mMS | At Week 64
  Endoscopic improvement defined as MES ≤ 1
PK Lead-In Cohort 2: Achievement of endoscopic improvement among Week 12 responders per mMS | At Week 64
  Endoscopic improvement defined as MES ≤ 1
PK Lead-In Cohort 1: Ability to discontinue corticosteroids prior to Week 64 (at least 90 days without corticosteroid exposure) and achievement of clinical remission per mMS among Week 12 responders per mMS | Up to Week 64
PK Lead-In Cohort 2: Ability to discontinue corticosteroids prior to Week 64 (at least 90 days without corticosteroid exposure) and achievement of clinical remission per mMS among Week 12 responders per mMS | Up to Week 64
Expansion Cohort 3: Achievement of clinical remission per mMS | At Week 12
Expansion Cohort 3: Achievement of clinical response per mMS | At Week 12
Expansion Cohort 3: Achievement of endoscopic improvement | At Week 12
Expansion Cohort 3: Symptomatic response per partial mMS | At Week 12
Expansion Cohort 3: Achievement of clinical response per mMS among Week 12 responders per mMS | At Week 64
Expansion Cohort 3: Achievement of endoscopic improvement among Week 12 responders per mMS | At Week 64
Expansion Cohort 3: Achievement of corticosteroid-free clinical remission per mMS among Week 12 responders per mMS | At Week 64

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (33):
- United States (6):
  - Phoenix Children's Hospital /ID# 273015, Phoenix, Arizona
  - Nicklaus Children'S Hospital - Miami - Southwest 62nd Avenue /ID# 271585, Miami, Florida
  - Childrens Center For Digestive Health Care /ID# 273228, Atlanta, Georgia
  - Goryeb Children's Hospital /ID# 271801, Morristown, New Jersey
  - Upmc Children'S Hospital Of Pittsburgh /ID# 272328, Pittsburgh, Pennsylvania
  - Patewood Medical Campus /ID# 272477, Greenville, South Carolina
- Belgium (3):
  - Cliniques Universitaires UCL Saint-Luc /ID# 270123, Brussels, Brussels Capital
  - Centre Hospitalier Régional de la Citadelle /ID# 270459, Liège, Liege
  - Hospital Universite Enfants Reine Fabiola /ID# 271860, Brussels
- Germany (3):
  - Medizinische Universitaet Lausitz - Carl Thiem /ID# 272023, Cottbus, Brandenburg
  - Klinikum Kassel /ID# 271546, Kassel, Hesse
  - Universitaetsklinikum Muenster /ID# 271898, Münster, North Rhine-Westphalia
- Greece (3):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 270143, Athens, Attica
  - University General Hospital Attikon /ID# 272361, Athens, Attica
  - General Hospital of Thessaloniki Hippokrateio /ID# 271939, Thessaloniki
- Italy (4):
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 271889, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Federico II /ID# 271895, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 272967, Rome, Roma
  - Ospedale Infantile Burlo Garofolo /ID# 274442, Trieste
- Serbia (3):
  - University Children's Hospital /ID# 269960, Belgrade, Beograd
  - Institut za zdravstvenu zastitu majke i deteta Srbije Dr Vukan Cupic /ID# 270696, Belgrade-Vračar, Beograd
  - Institute for Child and Youth Health Care of Vojvodina /ID# 269961, Novi Sad
- South Korea (5):
  - Pusan National University Yangsan Hospital /ID# 272769, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital /ID# 272852, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 273333, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 272894, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 272862, Seoul, Seoul Teugbyeolsi
- Spain (2):
  - Hospital Teresa Herrera - CHUAC /ID# 271459, A Coruña, A Coruna
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 271466, Majadahonda, Madrid
- Sweden (2):
  - Sodersjukhuset /ID# 271678, Stockholm, Stockholm County
  - Sahlgrenska Universitetssjukhuset /ID# 271675, Gothenburg, Västra Götaland County
- Taiwan (2):
  - Taichung Veterans General Hospital /ID# 269242, Taichung
  - National Taiwan University Hospital /ID# 269244, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com